CLINICAL TRIAL: NCT06635096
Title: A Prospective, Single-center, Single-arm Phase II Clinical Trial to Evaluate the Safety and Efficacy of Multimodal Thermal Therapy in the Treatment of Early-stage Invasive Breast Cancer
Brief Title: The Safety and Efficacy of Multimodal Thermal Therapy in the Treatment of Early-stage Invasive Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Director of General Surgery of Fudan Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTT-BC-001
Record Dates: First submitted 2024-09-25; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Thermal Therapy alone (Experimental): Multimodal Thermal Therapy
  Interventions: Device: Multimodal Tumor Thermal Therapy System (Shanghai MAaGI Medical Technology Co., Ltd.)

INTERVENTIONS:
Device: Multimodal Tumor Thermal Therapy System (Shanghai MAaGI Medical Technology Co., Ltd.) — These patients will receive multimodal thermal therapy using Multimodal Tumor Thermal Therapy System.

SUMMARY:
Multimodal thermal therapy (MTT), as an initiative integration of cryotherapy and radiofrequency heating, has been applied to treat various solid tumors. However, the feasibility and safety for MTT in the treatment of breast cancer is unknown. This prospective, open-label, single-arm phase II clinical study aimed to evaluate the efficacy and safety of MTT in the treatment of early-stage invasive breast cancer, and to explore the ablation-induced immune activating response.

ELIGIBILITY:
Inclusion Criteria:

1. Female，age 18-80 years.
2. Invasive carcinoma confirmed by core biopsy.
3. Newly diagnosed breast cancer patients, without neoadjuvant therapy.
4. Imaging findings showed an unifocal breast tumor with a maximum diameter of 2 cm, with no distant metastasis, no calcification, no skin or nipple adhesion, and no invasion of chest wall.
5. The functional level of major organs must meet the following requirements: blood routine: neutrophil (ANC)≥1.5×10^9/L; platelet count (PLT) ≥ (PLT)≥90×10^9/L; hemoglobin (Hb) ≥90g/L; coagulation: international normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5×ULN.

Exclusion Criteria:

1. Tumor involving skin, ulceration, inflammatory breast cancer patients.
2. Tumor involving the superficial layer of the skin.
3. KPS score < 70, or ECOG score > 2
4. Prior radiotherapy or prior use of investigational drugs or other immunosuppressive agents.
5. Heart, brain, lung, kidney and other vital organ failure.
6. Uncorrectable severe coagulopathy
7. Patient is pregnant or lactating
8. Poor glycemic control in diabetes
9. Patients with foreign body implantation around the tumor (such as breast augmentation injections or prostheses).
10. Patients with severe scars on the skin of the treatment area (protruding from the skin surface, width ≥ 1 cm)
11. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B indicates antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection of the analytical method).
12. Concurrent medical conditions that, in the judgment of the investigator, would jeopardize the subject's safety, could confound the study results, or affect the subject's completion of this study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-08 (Estimated); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate | 3 months
  The complete ablation rate was confirmed by core needle biopsy 3 months after multimodal thermal therapy. Complete ablation was defined as: tissue section at the ablation margin that was negative by histochemical staining.

SECONDARY OUTCOMES:
Safety of Multimodal Tumor Thermal Therapy | In 1 year
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0.
Breast MRI confirmed complete ablation. | In 6 months
  According to the mRECIST criteria, the complete ablation was confirmed by breast MRI in 6 months after multimodal thermal therapy.
Breast self evaluation | In 1 year
  Breast self evaluation for patients will be assessed by Functional Assessment of Cancer Therapy - Breast (FACT-B) scale scores.The FACT-B consists of 44 self-report items and assesses the specific breast cancer-related quality of life on 4 general and 1 breast-cancer specific subscale. A higher score indicates a higher cancer-related quality of life.
Assessment of immune activating response | In 1 year
  Immune indicator analysis will be conducted to evaluate the immune status and response of participants to the intervention. This will include the assessment of various immune cell populations and markers, such as:
  * CD4+ and CD8+ T lymphocyte counts and ratios.
  * B cell counts and subsets.
  * Dendritic cell (DC) counts and functionality.
  * Monocyte counts and subsets.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China